CLINICAL TRIAL: NCT02444858
Title: Safety and Efficacy of Human Umbilical-Cord-derived Mesenchymal Stem Cell Transplantation in Paraquat Poisoning Induced Lung Injury
Brief Title: Human Umbilical-Cord-Derived Mesenchymal Stem Cell Therapy in Paraquat Poisoning Induced Lung Injury
Acronym: UCMSC-PQLI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Ivy Institute of Stem Cells Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307-IVY-SC-004
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Paraquat Poisoning; Lung Injury
Keywords: paraquat poisoning; lung injury; stem cell therapy; human umbilical cord mesenchymal stem cell; phase 1/2 clinical study; allogeneic stem cell transplantation
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSC group (Experimental): Human umbilical cord MSCs are administrated to patients by intravenous injection
  Interventions: Biological: UCMSC group
- Control group(Normal saline) (Other): Patients will receive normal saline at the same time points as that in experimental group.
  Interventions: Other: Control group(Normal saline)

INTERVENTIONS:
Biological: UCMSC group — Human umbilical cord MSCs are transplanted by intravenous injection(5×10^5/kg) ，once a day,a total of three times.
  Arms: UCMSC group
Other: Control group(Normal saline) — Normal saline in same volume as MSCs are transplanted to patients.
  Arms: Control group(Normal saline)

SUMMARY:
Phase I-II Clinical Trial-Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with paraquat poisoning induced lung injury, randomized,single blind, controlled prospective study.

DETAILED DESCRIPTION:
Phase I-II Clinical Trial-Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with paraquat poisoning induced lung injury,randomized, single blind, controlled prospective study.

Forty patients will be selected and randomized into two groups: the first group of 20 patients will receive three-time injection of UC-MSC and the remaining 20 patients will comprise the control group.

Every patient will maintain their standard treatment of paraquat poisoning, with maximum tolerated dosage without side effects.

The day of last infusion will be considered day zero. From that moment, followup will be divided into 2 d,7 d,14 d, 28 d and 2 m.

Clinical results will be analyzed after completion of 2 months of followup.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 60 y(including 15y)
* A history of ingestion paraquat, and hospitalization within 96 hours after paraquat poisoning
* No previous organic disease history of serious heart, liver, kidney and lung, etc;
* Patients with moderate poisoning (oral dose of 20-40mg of PQ ion/kg of body weight)
* Patient or his legal agent signed informed consent voluntarily
* Capable of good communication with researchers and follow the entire test requirements

Exclusion Criteria:

* Refused to sign informed consent
* Elderly high-risk patients
* Socially and mentally disabilities
* Hepatitis B, hepatitis C, HIV and tuberculosis patients
* Pregnant or perinatal women
* Severe organ failure patients
* Patients participated in clinical trials of other drugs within 3 months
* Other circumstances not suitable to the trial(mixed toxicants poisoning)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety will be determined by the assessment of major adverse events. | 2 months
  Safety will be determined by the assessment of major adverse events defined as trial-related death,required hospitalization or prolonged hospitalization time, persistent or significant loss of organ function，other serious adverse events.

SECONDARY OUTCOMES:
The efficacy of UC-MSC treatment was measured clinical evaluation. | 2 months
  The efficacy of UC-MSC treatment was measured clinical evaluation defined as wheezing, coughing and other symptoms improved than before.
The efficacy of UC-MSC treatment was measured by chest computerized tomography. | 2 months
  The efficacy of UC-MSC treatment was quantified by the differences between the two groups and from baseline to 2 months, as measured by chest computerized tomography(CT).
The efficacy of UC-MSC treatment was monitored by pulmonary function. | 2 months
  The pulmonary function efficacy of UC-MSC treatment was measured by arterial blood gas analysis (oxygenation index).
The efficacy of UC-MSC treatment was measured by lab Indicators. | 2 months
  The efficacy of UC-MSC treatment was measured by lab Indicators defined as blood cell analysis, markers of inflammation (C-reactive protein).

CONTACTS AND LOCATIONS:
Overall Officials: Bing Liu, M.D., Study Chair — 307-IVY Translational Medicine Center; Zewu Qiu, M.D., Study Director — Department of poisoning treatment,Affiliated Hospital to Academy of Military Medical Sciences; Haochun Wang, M.D., Principal Investigator — Department of poisoning treatment,Affiliated Hospital to Academy of Military Medical Sciences; Xiaobo Peng, M.D., Principal Investigator — Department of poisoning treatment,Affiliated Hospital to Academy of Military Medical Sciences; Chunyan Wang, M.D., Principal Investigator — Department of poisoning treatment,Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of poisoning and treatment,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China